CLINICAL TRIAL: NCT06590675
Title: Development and Evaluation of a ChlorHexidine Gluconate bAthing pRotocol for Healthcare Settings in Low- and Middle-income Countries
Acronym: CHARM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding Withdrawn
Sponsor: University of Pennsylvania (Other)
Collaborators: Children's Hospital of Philadelphia (Other); University of Botswana (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); University of Utah (Other); Imperial College London (Other); Botswana-UPenn Partnership (Other)
Responsible Party: Principal Investigator, Ebbing Lautenbach, Principal Investigator, University of Pennsylvania
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 855362
Record Dates: First submitted 2024-05-29; First posted 2024-09-19 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Multidrug Resistant Bacterial Infection
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Intervention Model Description: This is a mixed methods study involving both a prospective interventional cohort study following approximately 240 neonates, and qualitative interviews of 10 caregivers and 20 healthcare workers in the neonatal unit (NNU) and intensive care unit (ICU).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ≥34 Week Neonates & ≥1.4 kg (Experimental): Phase 1 of a step-wise enrollment strategy in which chlorhexidine gluconate (CHG) bathing will be administered as follows:
  1. 1% CHG administered twice (2) a week (N=10)
  2. 1% CHG administered five times (5) a week (N=10)
  3. 2% CHG administered twice (2) a week (N=10)
  4. 2% CHG administered five times (5) a week (N=10)
  Interventions: Drug: Chlorhexidine Gluconate (CHG)
- ≥32 Week Neonates &/or 1.2 kg - 1.4 kg (Experimental): Phase 2 of a step-wise enrollment strategy in which chlorhexidine gluconate (CHG) bathing will be administered as follows:
  1. 1% CHG administered twice (2) a week (N=20)
  2. 1% CHG administered five times (5) a week (N=20)
  3. 2% CHG administered twice (2) a week (N=20)
  4. 2% CHG administered five times (5) a week (N=20)
  Interventions: Drug: Chlorhexidine Gluconate (CHG)
- ≥28 Week Neonates &/or 1.0 kg - 1.2 kg (Experimental): Phase 3 of a step-wise enrollment strategy in which chlorhexidine gluconate (CHG) bathing will be administered as follows:
  1. 1% CHG administered twice (2) a week (N=30)
  2. 1% CHG administered five times (5) a week (N=30)
  3. 2% CHG administered twice (2) a week (N=30)
  4. 2% CHG administered five times (5) a week (N=20)
  Interventions: Drug: Chlorhexidine Gluconate (CHG)
- Feasibility Assessment (No Intervention): Semi-structured, qualitative Interviews will be performed with caregivers (N=10) of neonates enrolled in the interventional arms and with healthcare workers (N=20) who care for these neonates in the neonatal unit (NNU) and intensive care unit (ICU).

INTERVENTIONS:
Drug: Chlorhexidine Gluconate (CHG) — A locally-prepared CHG formulation as a 1% or 2% solution
  Other Names: Aqueous CHG
  Arms: ≥28 Week Neonates &/or 1.0 kg - 1.2 kg; ≥32 Week Neonates &/or 1.2 kg - 1.4 kg; ≥34 Week Neonates & ≥1.4 kg

SUMMARY:
The overall goal of the ChlorHexidine gluconate (CHG) bAthing pRotocol for healthcare settings in low- and Middle-income countries (CHARM) study is to explore the safety, efficacy and feasibility of utilizing a locally prepared CHG solution and bathing protocol among hospitalized neonates to reduce bacterial colonization and healthcare-associated infection (HAI) burden in hospitalized patients.

DETAILED DESCRIPTION:
Neonatal sepsis is the third most common cause of neonatal deaths and multidrug-resistant Gram-negative bacteria are now the leading cause of sepsis among hospitalized neonates in south Asia and sub-Saharan Africa, including Botswana. Multidrug-Resistant Organism (MDRO) colonization is thought to precede infection, meaning that pathogens usually are transferred to the skin or intestinal mucosa where they live prior to translocating to the bloodstream or other sterile body compartments, triggering an inflammatory response recognized as clinical sepsis. Colonization is established through direct or indirect contact between a patient and a reservoir that harbors the pathogen.

Multidisciplinary infection prevention and control (IPC) practices can reduce the risk of neonatal MDRO colonization, but once colonized, newborns run the risk of acquiring a serious infection with a difficult-to-treat organism. The use of ancillary IPC measures, including chlorhexidine gluconate (CHG) bathing, has been studied as a de-colonization measure among hospitalized patients. CHG bathing is widely used in Intensive Care Units (ICUs) across high-income countries to reduce bacterial colonization with pathogens, and is being used more frequently in Neonatal Units (NNUs) in low and middle-income countries (LMICs) as a sepsis prevention measure.

The investigators of the CHARM study have developed a protocol to accomplish the following goals:

1. develop a low-cost, standardized protocol for CHG bathing in the ICU and NNU
2. assess safety of local CHG preparation among hospitalized neonates
3. determine the efficacy of CHG bathing using the developed protocol to reduce bacterial colonization and healthcare-associated infection (HAI) burden in hospitalized patients
4. to assess the feasibility and acceptability of CHG bathing among staff and caregivers

The investigators will utilize a mixed methods study involving both a prospective interventional cohort study following approximately 240 neonates, and qualitative interviews of 10 caregivers and 20 healthcare workers in the NNU and ICU.

ELIGIBILITY:
Inclusion Criteria:

* Neonates 1-6 days old admitted to the neo-natal unit expected to stay at least 7 days

Exclusion Criteria:

* Patients with a current weight of <1kg
* Patients with a current corrected gestational age of <28 weeks (by Ballard score, or by dates if Ballard is not done)
* Patients with a current diagnosis of hypothermia
* Patients with a current diagnosis of skin rash or skin injury

Ages: 1 Day to 6 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2025-02-19 (Actual); Primary Completion 2025-03-19 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Safety of locally prepared 1% and 2% chlorhexidine gluconate (CHG) cleansing: Skin integrity | At baseline and 30 minutes post application of CHG solution
  Skin condition score: Assessing skin reactions in neonates by a trained study nurse using the Darmstadt scale. The skin of the neonate will be assessed using a scale of 1 to 9, with 1 being the best condition and 9 being the worst condition, based on the following variables: skin breakdown, skin dryness, and erythema.
  Stopping rule: Skin fissuring (skin score of >3)
Safety of locally prepared 1% and 2% CHG cleansing: Systemic responses | At baseline and 30 minutes post application of CHG solution
  Temperature assessments will be performed at baseline and 30 min after application. If hypothermia is detected (defined as temperature below 36.5 C when measured from the same site at 30 minutes), the baby will be bundled and temperature retaken after 30 additional minutes. Babies will also be observed for 30 min for signs of anaphylaxis. Respiratory distress, cyanosis, urticaria, edema, vomiting/diarrhea, or lethargy will elicit a full set of vital signs to assess for hypotension and tachycardia.
  Stopping rule: Anaphylaxis, or any other rapid decompensation not explained by a patient's concurrent conditions

SECONDARY OUTCOMES:
Reduction in pathogen colonization of participants receiving CHG cleansing: -1% vs 2% CHG -2x vs 5x weekly frequency | 2x/week cleansing within 96 hours after last CHG application; 5x/week cleansing within 72 hours after last CHG application
  Trained research personnel will use flocked swabs to collect perirectal and umbilical swabs. For perirectal samples, the swab tip will be gently introduced around the anus. For skin samples, a single swab will be rubbed back-and-forth around the umbilicus. All swabs collected from neonates will be placed into transport media. The samples will be labeled with the infant's study number, source of sample and timing of sample.
  At the National Health Laboratory microbiology section, swab specimens will be directly inoculated on chromogenic culture media which is selective and differential for select multidrug-resistant organisms (MDROs). MDRO isolates will then undergo confirmatory identification and sensitivity testing using the VITEK® 2 platform. Results will be available within 72 hrs of delivery to the laboratory.
Reduction in bloodstream infection of participants receiving CHG cleansing: -1% vs 2% CHG -2x vs 5x weekly frequency | Within 30 days of initiating CHG intervention
  Blood culture surveillance data will be extracted to determine incidence of blood stream infection within 30 days of initiating CHG intervention by enrollment band both ward-level and among study participants, stratified by weight/gestational age.

CONTACTS AND LOCATIONS:
Overall Officials: Ebbing Lautenbach, MD,MPH,MSCE, Principal Investigator — University of Pennsylvania; Susan Coffin, MD,MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gezmu AM, Bulabula ANH, Dramowski A, Bekker A, Aucamp M, Souda S, Nakstad B. Laboratory-confirmed bloodstream infections in two large neonatal units in sub-Saharan Africa. Int J Infect Dis. 2021 Feb;103:201-207. doi: 10.1016/j.ijid.2020.11.169. Epub 2020 Nov 20. PMID 33227511
- [Background] Kabwe M, Tembo J, Chilukutu L, Chilufya M, Ngulube F, Lukwesa C, Kapasa M, Enne V, Wexner H, Mwananyanda L, Hamer DH, Sinyangwe S, Ahmed Y, Klein N, Maeurer M, Zumla A, Bates M. Etiology, Antibiotic Resistance and Risk Factors for Neonatal Sepsis in a Large Referral Center in Zambia. Pediatr Infect Dis J. 2016 Jul;35(7):e191-8. doi: 10.1097/INF.0000000000001154. PMID 27031259
- [Background] Flokas ME, Karanika S, Alevizakos M, Mylonakis E. Prevalence of ESBL-Producing Enterobacteriaceae in Pediatric Bloodstream Infections: A Systematic Review and Meta-Analysis. PLoS One. 2017 Jan 31;12(1):e0171216. doi: 10.1371/journal.pone.0171216. eCollection 2017. PMID 28141845
- [Background] Strysko J, Machiya T, Lechiile K, et al. Carbapenem-resistant Acinetobacter baumannii at a tertiary-care hospital in Botswana: Focus on perinatal environmental exposures. (2022). Antimicrobial Stewardship & Healthcare Epidemiology, 2(S1), S79-S79. doi:10.1017/ash.2022.206
- [Background] Kagia N, Kosgei P, Ooko M, Wafula L, Mturi N, Anampiu K, Mwarumba S, Njuguna P, Seale AC, Berkley JA, Bottomley C, Scott JAG, Morpeth SC. Carriage and Acquisition of Extended-spectrum beta-Lactamase-producing Enterobacterales Among Neonates Admitted to Hospital in Kilifi, Kenya. Clin Infect Dis. 2019 Aug 16;69(5):751-759. doi: 10.1093/cid/ciy976. PMID 30830952
- [Background] Mwananyanda L, Pierre C, Mwansa J, Cowden C, Localio AR, Kapasa ML, Machona S, Musyani CL, Chilufya MM, Munanjala G, Lyondo A, Bates MA, Coffin SE, Hamer DH. Preventing Bloodstream Infections and Death in Zambian Neonates: Impact of a Low-cost Infection Control Bundle. Clin Infect Dis. 2019 Sep 27;69(8):1360-1367. doi: 10.1093/cid/ciy1114. PMID 30596901
- [Background] Dramowski A, Pillay S, Bekker A, Abrahams I, Cotton MF, Coffin SE, Whitelaw AC. Impact of 1% chlorhexidine gluconate bathing and emollient application on bacterial pathogen colonization dynamics in hospitalized preterm neonates - A pilot clinical trial. EClinicalMedicine. 2021 Jun 18;37:100946. doi: 10.1016/j.eclinm.2021.100946. eCollection 2021 Jul. PMID 34195575
- [Background] Musuuza JS, Roberts TJ, Hundt AS, Carayon P, Zimbric ML, Schuetz V, Reppen M, Smith W, Koffarnus K, Brown RL, Bowling J, Jalali K, Safdar N. Implementing daily chlorhexidine gluconate treatment for the prevention of healthcare-associated infections in non-intensive care settings: A multiple case analysis. PLoS One. 2020 Apr 24;15(4):e0232062. doi: 10.1371/journal.pone.0232062. eCollection 2020. PMID 32330165
- [Background] Silvestri DL, McEnery-Stonelake M. Chlorhexidine: uses and adverse reactions. Dermatitis. 2013 May-Jun;24(3):112-8. doi: 10.1097/DER.0b013e3182905561. PMID 23665831
- [Background] Garland JS, Alex CP, Mueller CD, Otten D, Shivpuri C, Harris MC, Naples M, Pellegrini J, Buck RK, McAuliffe TL, Goldmann DA, Maki DG. A randomized trial comparing povidone-iodine to a chlorhexidine gluconate-impregnated dressing for prevention of central venous catheter infections in neonates. Pediatrics. 2001 Jun;107(6):1431-6. doi: 10.1542/peds.107.6.1431. PMID 11389271
- [Background] Visscher M, deCastro MV, Combs L, Perkins L, Winer J, Schwegman N, Burkhart C, Bondurant P. Effect of chlorhexidine gluconate on the skin integrity at PICC line sites. J Perinatol. 2009 Dec;29(12):802-7. doi: 10.1038/jp.2009.116. Epub 2009 Aug 20. PMID 19693022
- [Background] Darmstadt GL, Badrawi N, Law PA, Ahmed S, Bashir M, Iskander I, Al Said D, El Kholy A, Husein MH, Alam A, Winch PJ, Gipson R, Santosham M. Topically applied sunflower seed oil prevents invasive bacterial infections in preterm infants in Egypt: a randomized, controlled clinical trial. Pediatr Infect Dis J. 2004 Aug;23(8):719-25. doi: 10.1097/01.inf.0000133047.50836.6f. PMID 15295221
- [Background] Mullany LC, Khatry SK, Sherchand JB, LeClerq SC, Darmstadt GL, Katz J, Gauchan P, Adhikari RK, Rana A, Tielsch JM. A randomized controlled trial of the impact of chlorhexidine skin cleansing on bacterial colonization of hospital-born infants in Nepal. Pediatr Infect Dis J. 2008 Jun;27(6):505-11. doi: 10.1097/INF.0b013e31816791a2. PMID 18449064
- [Background] Krautheim AB, Jermann TH, Bircher AJ. Chlorhexidine anaphylaxis: case report and review of the literature. Contact Dermatitis. 2004 Mar;50(3):113-6. doi: 10.1111/j.0105-1873.2004.00308.x. PMID 15153122